CLINICAL TRIAL: NCT02627183
Title: Circulating Brain-derived Neurotrophic Factor (BDNF) in Patients With Atrial Fibrillation Undergoing Catheter Ablation or Exercise Training: A Pilot Study (NEURO-AF)
Brief Title: Circulating BDNF in Patients With Atrial Fibrillation Undergoing Catheter Ablation or Exercise Training
Acronym: NEURO-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 20150742
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Paroxysmal AF + catheter ablation: Subjects with paroxysmal Atrial Fibrillation (AF) undergoing catheter ablation.
  Interventions: Procedure: Catheter ablation
- Permanent/persistent AF + exercise: Subjects with permanent or persistent Atrial Fibrillation (AF) undergoing exercise training two times weekly for 12 weeks as part of their involvement in the OPPORTUNITY Study (NCT02602457).
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Procedure: Catheter ablation — Subjects undergoing catheter ablation for the first time for atrial fibrillation as part of their regular care (regardless of involvement in this study).
  Groups: Paroxysmal AF + catheter ablation
Behavioral: Exercise training — Subjects participating in supervised exercise classes for up to 60 minutes in length 2 times/week as part of their involvement in another study (NCT02602457).
  Groups: Permanent/persistent AF + exercise

SUMMARY:
The main purpose of this project is to determine the impact of atrial fibrillation interventions (catheter ablation and exercise training) on circulating BDNF concentrations in patients with atrial fibrillation. It also seeks to determine if there is a relation between circulating BDNF concentrations and mental health (depression severity, quality of life and symptoms) among those undergoing interventions for atrial fibrillation catheter ablation or exercise training.

DETAILED DESCRIPTION:
The main purpose of this project is to determine the impact of atrial fibrillation interventions (catheter ablation and exercise training) on circulating BDNF concentrations in patients with atrial fibrillation. It also seeks to determine if there is a relation between circulating BDNF concentrations and mental health (depression severity, quality of life and symptoms) among those undergoing interventions for atrial fibrillation catheter ablation or exercise training. Using a pre-post study design, the investigators will explore interventions in two subsets of patients at the opposite end of the atrial fibrillation clinical spectrum. Arm 1: patients with paroxysmal atrial fibrillation will undergo catheter ablation (n=100). Arm 2: patients with permanent or persistent atrial fibrillation will perform exercise training 2 times weekly for 12 weeks (n=100). Total sample size will be 200 participants. All measurements will be performed at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be either currently enrolled in the OPPORTUNITY trial (NCT02602457) or have paroxysmal atrial fibrillation and be scheduled to undergo catheter ablation (for the first time) through the electrophysiology clinic at the University of Ottawa Heart Institute.
2. Subjects must be willing and able to provide a blood sample.
3. Subjects must be willing and able to provide informed consent.

Exclusion Criteria:

1. Subject is not either currently enrolled in the OPPORTUNITY trial (NCT02602457) or scheduled to undergo catheter ablation (for the first time) through the electrophysiology clinic at the University of Ottawa Heart Institute for paroxysmal atrial fibrillation.
2. Subjects with congestive heart failure with heart failure admission in the past 3 months.
3. Subjects with a cerebrovascular accident in the past 3 months
4. Subjects with severe dementia.
5. Subjects with a history of severe psychiatric illness (e.g., schizoaffective disorder, bipolar disorder, or schizophrenia).
6. Subjects with an active infection or inflammatory condition.
7. Subjects who are pregnant, lactating or planning to become pregnant during the study period.
8. Subject is unable to read or understand English or French.
9. Subject is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with paroxysmal atrial fibrillation that will undergo catheter ablation and subjects with permanent or persistent atrial fibrillation undergoing exercise training two times weekly for 12 weeks as part of their involvement in the OPPORTUNITY Study (NCT02602457).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Changes in circulating BDNF concentrations measured by blood samples collected from subjects with atrial fibrillation | approximately 3 months post catheter ablation or following the 12 week exercise training intervention period
  Changes in circulating BDNF concentrations measured by blood samples collected from subjects with atrial fibrillation approximately 3 months post catheter ablation or following the 12 week exercise training intervention.

SECONDARY OUTCOMES:
Changes in subjects' symptoms measured by the patient diary for symptoms | approximately 3 months post catheter ablation or following the 12 week exercise training intervention period
  Changes in subjects' symptoms measured by the patient diary for symptoms approximately 3 months post catheter ablation or following the 12 week exercise training intervention period.
Changes in depression severity measured using the Beck Depression Inventory II (BDI-II) | approximately 3 months post catheter ablation or following the 12 week exercise training intervention period
  Changes in depression severity measured using the Beck Depression Inventory II (BDI-II) approximately 3 months after catheter ablation or following the 12 week exercise training intervention period.
Changes in general quality of life as measured by the Short Form Health Survey 36 (SF-36) | approximately 3 months post catheter ablation or following the 12 week exercise training intervention period
  Changes in general quality of life as measured by the Short Form Health Survey 36 (SF-36) approximately 3 months after catheter ablation or following the 12 week exercise training intervention period.
Changes in disease specific quality of life measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS) | approximately 3 months post catheter ablation or following the 12 week exercise training intervention period
  Changes in disease specific quality of life measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS) approximately 3 months after catheter ablation or following the 12 week exercise training intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Girish Nair, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada